CLINICAL TRIAL: NCT00460109
Title: A Phase II Clinical Trial of Denileukin Diftitox in Combination With Rituximab in Previously Untreated Follicular B-Cell Non-Hodgkin's Lymphoma
Brief Title: Rituximab and Denileukin Diftitox in Treating Patients With Previously Untreated Stage III or Stage IV Follicular B-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0682; NCI-2009-00662 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000539551 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — denileukin diftitox; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rituximab + denileukin diftitox (Experimental): Patients receive rituximab IV on days 1, 8, 15, and 22. Patients also receive denileukin diftitox IV over 15-60 minutes on days 1-5. Treatment with denileukin diftitox repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: denileukin diftitox; Biological: rituximab

INTERVENTIONS:
Biological: denileukin diftitox
Biological: rituximab

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Combinations of biological substances in denileukin diftitox may be able to carry cancer-killing substances directly to cancer cells. Giving rituximab together with denileukin diftitox may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving rituximab together with denileukin diftitox works in treating patients with previously untreated stage III or stage IV follicular B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate (complete response [CR], unconfirmed CR, and partial response) in patients with previously untreated stage III or IV follicular B-cell non-Hodgkin's lymphoma treated with rituximab and denileukin diftitox.
* Assess the overall survival, time-to-progression, duration of response, and time-to-new therapy in patients treated with this regimen.

Secondary

* Determine whether this regimen depletes or inhibits the function of regulatory T cells in these patients.

OUTLINE: This is a multicenter study.

Patients receive rituximab IV on days 1, 8, 15, and 22. Patients also receive denileukin diftitox IV over 15-60 minutes on days 1-5. Treatment with denileukin diftitox repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Blood is collected at baseline; on day 1 of courses 2-4; and 1 and 4 months after completion of study treatment for research studies. Research studies include analysis of peripheral blood lymphocyte subsets expressing CD3, CD4, CD8, CD19, CD25, and CD26 by flow cytometry; quantitation of CD4+, CD25+ regulatory T cells by flow cytometry; tumor-specific γ-interferon-secreting T cells by enzyme-linked immunospot assay; tumor-specific cytotoxic T-lymphocyte activity; and immune activation by enzyme-linked immunosorbent assay.

After completion of study treatment, patients are followed periodically for up to 5 years after registration.

PROJECTED ACCRUAL: A total of 53 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed follicular B-cell non-Hodgkin's lymphoma (NHL)

  * Stage III or IV disease
  * Grade 1 or 2 disease
* Previously untreated disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques

  * Clearly defined bidimensional diameter ≥ 2 x 2 cm on physical examination OR > 2.0 cm in 1 of the dimensions by CT scan, MRI, or plain radiograph imaging
  * Splenic enlargement may be used as a measurable parameter if the spleen is palpable ≥ 3 cm below the left costal margin
* Circulating tumor cells < 5,000/mm³
* Must have paraffin-embedded tissue blocks/slides available
* No CNS lymphoma

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 1 year
* WBC ≥ 3,400/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10.0 g/dL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 times ULN
* AST ≤ 3 times ULN
* Creatinine ≤ 1.5 times ULN
* Albumin ≥ 3 g/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 year after completion of study therapy
* No HIV infection
* No other active malignancies
* No active uncontrolled infection
* No known hypersensitivity to denileukin diftitox or any of its components, including diphtheria toxin, aldesleukin, or excipients

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, immunotherapy, vaccines, or radiotherapy for NHL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-04; Primary Completion 2010-10 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M. Ansell, MD, PhD, Study Chair — Mayo Clinic
Locations (165):
- United States (165):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Anthony's Memorial Hospital, Effingham, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls Medical Group, PA, Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Ansell SM, Tang H, Kurtin PJ, Koenig PA, Nowakowski GS, Nikcevich DA, Nelson GD, Yang Z, Grote DM, Ziesmer SC, Silberstein PT, Erlichman C, Witzig TE. Denileukin diftitox in combination with rituximab for previously untreated follicular B-cell non-Hodgkin's lymphoma. Leukemia. 2012 May;26(5):1046-52. doi: 10.1038/leu.2011.297. Epub 2011 Oct 21. PMID 22015775

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab + Denileukin Diftitox: Patients receive 375 mg/m^2 rituximab IV on days 1, 8, 15, and 22. Patients also receive 18 mcg/kg/day denileukin diftitox IV over 15-60 minutes on days 1-5. Treatment with denileukin diftitox repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Rituximab + Denileukin Diftitox
Started | 24
Completed | 23
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab + Denileukin Diftitox
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 60.0 [27.0 to 79.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Confirmed Tumor Response (Complete Response [CR], Unconfirmed CR, and Partial Response)
Description: A confirmed tumor response is defined to be either a CR, CRu or PR. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Response criteria for non-Hodgkin's lymphoma (NHL) will be followed. Complete response (CR): (a) Complete disappearance of all detectable disease and disease-related symptoms; (b) All lymph nodes and nodal masses must have regressed to normal size; (c) the spleen must have regressed; CR/unconfirmed (CRu): Those patients who fulfill the criteria in (a) and (c), but with a residual lymph node mass that has regressed by more that 75% in the sum of the products of the greatest diameters (SPD). Partial response (PR): ≥50% decrease in SPD of the six largest dominant nodes or nodal masses; no increase in the size of other nodes, liver, or spleen. Splenic and hepatic nodules must regress by at least 50% in the SPD; No new sites of disease.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Rituximab + Denileukin Diftitox
Number analyzed (Participants) | 23
proportion of participants | 0.48 [0.27 to 0.69]

2. Secondary Outcome: Survival Time
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval)
Arm/Group | Rituximab + Denileukin Diftitox
Number analyzed (Participants) | 23
Value | NA [NA to NA] — The median overall survival was not reached.

3. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the time from registration to the earliest date of documentation of disease progression. If a patient dies without a documentation of disease progression the patient will be considered to have had tumor progression at the time of their death unless there is sufficient documented evidence to conclude no progression occurred prior to death. The distribution of time to disease progression will be estimated using the method of Kaplan-Meier. Progression is defined using the response criteria for non-Hodgkin's lymphoma, as at least a 50% increase from nadir in the sum of the products of the greatest diameters (SPD) of any previously identified abnormal node for PRs or non-responders, or appearance of any new lesion during or at the end of therapy.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval)
Arm/Group | Rituximab + Denileukin Diftitox
Number analyzed (Participants) | 23
Value | NA [NA to NA] — Median time to progression was not reached.

4. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) is defined as the time from the date at which the patient's objective status is first noted to be either a CR, CRu or PR to the earliest date of progression. The distribution of DOR will be estimated using Kaplan-Meier methods. Response criteria for non-Hodgkin's lymphoma (NHL) will be followed. Complete response (CR): (a) Complete disappearance of all detectable disease and disease-related symptoms; (b) All lymph nodes and nodal masses must have regressed to normal size; (c) the spleen must have regressed; CR/unconfirmed (CRu): Those patients who fulfill the criteria in (a) and (c), but with a residual lymph node mass that has regressed by more that 75% in the sum of the products of the greatest diameters (SPD). Partial response (PR): ≥50% decrease in SPD of the six largest dominant nodes or nodal masses; no increase in the size of other nodes, liver, or spleen. Splenic and hepatic nodules must regress by at least 50% in the SPD; No new sites of disease.
Time Frame: Up to 5 years
Population: Overall Number of Participants Analyzed reflects only the number of participants with reported data for this outcome.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Denileukin Diftitox
Number analyzed (Participants) | 6
months | 22.5 [7.3 to 22.5]

5. Secondary Outcome: Time to Subsequent Therapy
Description: Time to subsequent therapy is defined to be the time from the end of active treatment date to the date subsequent therapy is initiated. The distribution of time to subsequent therapy will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Rituximab + Denileukin Diftitox
Number analyzed (Participants) | 23
months | NA [8.5 to NA] — Median Time to Subsequent Therapy and the upper limit of the 95% confidence interval were not reached.

ADVERSE EVENTS:
Time Frame: Adverse events are assessed during Treatment (weekly while receiving treatment and prior to the start of a new cycle) and during Observation (1 month after completing treatment, at 4, 7, and 10 months after completing treatment, 1 year after treatment, and every 6 months for years 2-5); up to 5 years.
Description: This study will utilize the Common Terminology Criteria for Adverse Events (CTCAE) v3.0 for adverse event monitoring and reporting. All graded adverse events are reported.
Arm/Group | Rituximab + Denileukin Diftitox
Serious Adverse Events (participants affected / at risk) | 7/23
Other Adverse Events (participants affected / at risk) | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab + Denileukin Diftitox (N=23)
Cardiac valve disease (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Premature ventricular contractions (Cardiac disorders) | 1 (1)
Ventricular bigeminy (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Localized edema (General disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1)
Creatine phosphokinase increased (Investigations) | 2 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 5 (5)
Hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab + Denileukin Diftitox (N=23)
Hemoglobin decreased (Blood and lymphatic system disorders) | 11 (26)
Cardiac pain (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Retinopathy (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 3 (3)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 3 (3)
Pain (General disorders) | 2 (2)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 6 (7)
Catheter related infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 6 (6)
Creatinine increased (Investigations) | 3 (3)
Laboratory test abnormal (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 3 (4)
Lymphocyte count decreased (Investigations) | 4 (4)
Neutrophil count decreased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 7 (8)
Blood glucose increased (Metabolism and nutrition disorders) | 4 (5)
Serum albumin decreased (Metabolism and nutrition disorders) | 9 (11)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Protein urine positive (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes